CLINICAL TRIAL: NCT05079074
Title: Clinical Application of Circulating Tumor DNA (ctDNA) to Monitor the Molecular Tumor Burden in Patients With Late-stage Breast Cancer
Brief Title: Clinical Application of Circulating Tumor DNA (ctDNA) in Patients With Late-stage Breast Cancer
Acronym: ACTDNA
Status: Completed | Type: Observational
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017YS031
Record Dates: First submitted 2021-09-23; First posted 2021-10-15 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Breast Cancer; Circulating Tumor DNA; Gene Abnormality
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peripheral blood lymphocytes (PBL) and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with late-stage metastatic breast cancers.: This cohort included patients with late-stage metastatic breast cancers and their disease progressed after at least two-line treatment.
  Interventions: Diagnostic Test: ctDNA testing

INTERVENTIONS:
Diagnostic Test: ctDNA testing — ctDNA testing was performed for late-stage metastatic breast cancer patients to trace their ctDNA abnormality.

SUMMARY:
This is a retrospective, observational, multi-center clinical study of circulating tumor DNA (ctDNA) application in late-stage breast cancers.

DETAILED DESCRIPTION:
This study aims to evaluate the feasibility of plasma ctDNA mutation spectrum and clonal spectrum in late-stage metastatic breast cancer patients. Meanwhile, this study tries to establish a model of ctDNA subtyping system to evaluate the molecular load of tumor, to evaluate the curative effect comprehensively and to detect the disease progression in advance. In addition, the investigators plan to explore the clonal evolution of ctDNA in patients with progressive disease (PD), and to monitor the changes of tumor heterogeneity from the molecular level, so as to provide reference for the analysis of drug sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Recent progression of TNBC after multiple lines of chemotherapy or of HR+ or HER2+ MBC after multiple lines of endocrine or targeted therapy;
* No available recommendation for the next treatment regimen;
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2;
* An updated, available pathological HR/HER2 status for metastasis;
* According to RECIST 1.1 standard, there should be at least one measurable target lesion;
* The expected survival time is > 3 months;
* Those aged 18-70 years old;
* Liver and kidney function and blood routine test meet the following conditions: Neutrophil > 2.0g/l, Hb > 9g / L, PLT > 100g / L; ALT and AST < 2.5ULN; TBIL < 1.5ULN; Cr < 1.0ULN
* Signing informed consent;
* Those willing to accept polygenic testing.

Exclusion Criteria:

* Patients with multiple primary tumors;
* Those who are unable to obtain blood samples;
* Those with a history of immunodeficiency or organ transplantation;
* Those with abnormal cardiac function or previous history of myocardial infarction or serious arrhythmia;
* The researchers think it is not suitable to participate in this experiment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cohort study recruited consecutive patients with recent progression of metastatic TNBC after multiple lines of chemotherapy or of HR+ or HER2+ metastatic breast cancer after multiple lines of endocrine or targeted therapy.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
ctDNA change index | From the date of recruitment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
  The dynamic change of the frequency spectrum of ctDNA mutation in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Quchang Ouyang, MD, Principal Investigator — Hunan Cancer Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crowley E, Di Nicolantonio F, Loupakis F, Bardelli A. Liquid biopsy: monitoring cancer-genetics in the blood. Nat Rev Clin Oncol. 2013 Aug;10(8):472-84. doi: 10.1038/nrclinonc.2013.110. Epub 2013 Jul 9. PMID 23836314
- [Background] Dawson SJ, Tsui DW, Murtaza M, Biggs H, Rueda OM, Chin SF, Dunning MJ, Gale D, Forshew T, Mahler-Araujo B, Rajan S, Humphray S, Becq J, Halsall D, Wallis M, Bentley D, Caldas C, Rosenfeld N. Analysis of circulating tumor DNA to monitor metastatic breast cancer. N Engl J Med. 2013 Mar 28;368(13):1199-209. doi: 10.1056/NEJMoa1213261. Epub 2013 Mar 13. PMID 23484797
- [Background] Garcia-Murillas I, Schiavon G, Weigelt B, Ng C, Hrebien S, Cutts RJ, Cheang M, Osin P, Nerurkar A, Kozarewa I, Garrido JA, Dowsett M, Reis-Filho JS, Smith IE, Turner NC. Mutation tracking in circulating tumor DNA predicts relapse in early breast cancer. Sci Transl Med. 2015 Aug 26;7(302):302ra133. doi: 10.1126/scitranslmed.aab0021. PMID 26311728
- [Background] Murtaza M, Dawson SJ, Pogrebniak K, Rueda OM, Provenzano E, Grant J, Chin SF, Tsui DWY, Marass F, Gale D, Ali HR, Shah P, Contente-Cuomo T, Farahani H, Shumansky K, Kingsbury Z, Humphray S, Bentley D, Shah SP, Wallis M, Rosenfeld N, Caldas C. Multifocal clonal evolution characterized using circulating tumour DNA in a case of metastatic breast cancer. Nat Commun. 2015 Nov 4;6:8760. doi: 10.1038/ncomms9760. PMID 26530965
- [Background] Swanton C, Govindan R. Clinical Implications of Genomic Discoveries in Lung Cancer. N Engl J Med. 2016 May 12;374(19):1864-73. doi: 10.1056/NEJMra1504688. No abstract available. PMID 27168435
- [Background] Yates LR, Gerstung M, Knappskog S, Desmedt C, Gundem G, Van Loo P, Aas T, Alexandrov LB, Larsimont D, Davies H, Li Y, Ju YS, Ramakrishna M, Haugland HK, Lilleng PK, Nik-Zainal S, McLaren S, Butler A, Martin S, Glodzik D, Menzies A, Raine K, Hinton J, Jones D, Mudie LJ, Jiang B, Vincent D, Greene-Colozzi A, Adnet PY, Fatima A, Maetens M, Ignatiadis M, Stratton MR, Sotiriou C, Richardson AL, Lonning PE, Wedge DC, Campbell PJ. Subclonal diversification of primary breast cancer revealed by multiregion sequencing. Nat Med. 2015 Jul;21(7):751-9. doi: 10.1038/nm.3886. Epub 2015 Jun 22. PMID 26099045
- [Result] Hu ZY, Xie N, Tian C, Yang X, Liu L, Li J, Xiao H, Wu H, Lu J, Gao J, Hu X, Cao M, Shui Z, Xiao M, Tang Y, He Q, Chang L, Xia X, Yi X, Liao Q, Ouyang Q. Identifying Circulating Tumor DNA Mutation Profiles in Metastatic Breast Cancer Patients with Multiline Resistance. EBioMedicine. 2018 Jun;32:111-118. doi: 10.1016/j.ebiom.2018.05.015. Epub 2018 May 26. PMID 29807833
- [Derived] Tang Y, Li J, Liu B, Ran J, Hu ZY, Ouyang Q. Circulating tumor DNA profile and its clinical significance in patients with hormone receptor-positive and HER2-negative mBC. Front Endocrinol (Lausanne). 2022 Nov 28;13:1075830. doi: 10.3389/fendo.2022.1075830. eCollection 2022. PMID 36518248
- [Derived] Hu ZY, Tang Y, Liu L, Xie N, Tian C, Liu B, Zou L, Zhou W, Wang Y, Xia X, Ouyang Q. Subtyping of metastatic breast cancer based on plasma circulating tumor DNA alterations: An observational, multicentre platform study. EClinicalMedicine. 2022 Jul 18;51:101567. doi: 10.1016/j.eclinm.2022.101567. eCollection 2022 Sep. PMID 35875816

DOCUMENTS (1):
  • Study Protocol (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT05079074/Prot_000.pdf